CLINICAL TRIAL: NCT06604052
Title: A Prospective, Randomized, Parallel-Controlled Study Comparing Laparoscopic/Robotic Stoma Reduced-Port Fusion Surgery with Traditional Surgery in Patients with Temporary Ileostomy
Brief Title: A Study Comparing Laparoscopic/Robotic Stoma Reduced-Port Fusion Surgery with Traditional Surgery in Patients with Temporary Ileostomy
Acronym: FUSION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Tingyu Wu, Principal Investigator, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XHEC-C-2024-158-2
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ileostomy
Keywords: ileostomy; minimally invasive surgery; Reduced-Port Fusion Surgery; stoma complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reduced-Port Fusion Surgery Group (Experimental): Recive preoperative trocar/stoma fusion positioning and intraoperative trocar/stoma fusion surgery
  Interventions: Procedure: Reduced-Port Fusion Surgery
- Traditional surgery group (Active Comparator): Recive traditional preoperative stoma positioning and traditional stoma surgery
  Interventions: Procedure: Traditional surgery

INTERVENTIONS:
Procedure: Reduced-Port Fusion Surgery — (1) The Joint Trocar/Stoma Zone will be delineated by the stoma therapist. (2) The placement of the fusion point will involve collaboration between the surgeon and stoma therapist. This will be based on the surgeon's trocar placement plan and the stoma therapist's positioning principles. (3) Follow the principles of modified stomal positioning. (4) The surgeon will insert the main trocar based on the preoperative positioning point. During stoma creation, the 12 mm main trocar incision will be extended to 25-30 mm to create an ileostomy.
  Arms: Reduced-Port Fusion Surgery Group
Procedure: Traditional surgery — (1) The stoma therapists perform stoma positioning using traditional stoma positioning method. The surgeon will determine the primary trocar location, ensuring it does not overlap with the stoma site. (2) The surgeon will insert the primary trocar based on the preoperative positioning point and conduct the surgery. During stoma creation, the surgeons create ileal stoma according to the preoperative stoma positioning point.
  Arms: Traditional surgery group

SUMMARY:
The traditional positioning and surgical methods for temporary ileostomy no longer meet the requirements of minimally invasive surgery: (1) Conventional stoma positioning often leads to the trocar incision being too close to the stoma site, increasing the risk of baseplate leakage and skin infection. (2) Since stoma positioning is required to be within the rectus abdominis, the proximity between the stoma and auxiliary incision can heighten difficulties in stoma bag attachment and raises the risk of fecal leakage. (3) Stoma retraction surgery within the rectus abdominis is more traumatic and complex. We introduce for the first time a modified stoma positioning and surgical method, termed Reduced-Port Fusion Surgery. This technique includes preoperative trocar/stoma fusion positioning and intraoperative trocar/stoma fusion surgery. The procedure is based on the 3R principles: Reposition - the stoma is repositioned within the Joint Trocar/Stoma Zone, allowing for more lateral placement to meet surgical needs without being confined to the rectus abdominis. Reduce Port - the same fusion point is used for both trocar insertion and stoma creation, enabling dual use of one site. Recognize - surgeons participate in stoma positioning, recognize the positioning, and follow the procedure. This prospective, randomized, parallel-controlled clinical study aims to evaluate whether Reduced-Port Fusion Surgery can reduce stoma-related complications, postoperative pain, improve quality of life, and facilitate stoma retraction surgery compared to traditional methods. A total of 80 participants will be randomly assigned in a 1:1 ratio. The experimental group will undergo Reduced-Port Fusion Surgery while the control group will receive traditional surgery.

ELIGIBILITY:
Inclusion Criteria:

1. After preoperative evaluation, patients scheduled for laparoscopic/robotic colorectal surgery (rectum, sigmoid colon, left colon) who are planned to undergo prophylactic ileostomy.
2. No serious systemic infection or immunosuppression.
3. Over 18 years of age.
4. Eastern Cooperative Oncology Group Performance Status: 0-1
5. The expected survival time > 6 months.
6. The subjects voluntarily participate and sign the informed consent

Exclusion Criteria:

1. Any skin infectious diseases in the abdominal wall.
2. Use hormones and immunosuppressive drugs within 1 month before surgery.
3. The time between operation and the last chemotherapy was less than 1 month.
4. Any previous ostomy surgery.
5. Any serious active infection or uncontrollable infection that requires systematic treatment.
6. A clear history of neurological or psychiatric disorders.
7. Subjects may not be able to complete the study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall complication rate of stoma | 7, 30, and 90 days after surgery
  Observe and assess for stoma complications

SECONDARY OUTCOMES:
DET（Discoloration，Erosion and Tissue overgrowth） score | 7, 30, and 90 days after surgery
  Measure the state of the skin around the stoma and the corresponding lesion area, ranging from 0-15, higher scores mean a worse outcome of stoma
Stomal skin infection rate | 7, 30, and 90 days after surgery
  Observe and assess for stomal skin infection rate
Parastostomy trocar incision infection rate | 7, 30, and 90 days after surgery
  To observe whether trocar incision infection occurred
Parastomal hernia rate | 7, 30, and 90 days after surgery
  To observe whether parastomal hernia occurred
Stoma Pain Score | 7, 30, and 90 days after surgery
  Measurement of stoma pain level using numerical rating scale，ranging from 0-10, higher scores mean a worse outcome of pain
Quality of life scale score | 30 and 90 days after surgery
  Measurement of quality of life for patients using the European Organization for Reasearch and Treatment of Cancer QLQ-C30 Questionnaire (EORTC QLQ-C30), ranging from 0-100, higher scores mean a better outcome of quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: Yes
In this study personal information and data such as patient history, physical examination results, surgical records, and study questionnaire data will be collected. These data will be used to evaluate the efficacy and safety of the new procedure and for academic publication. The researcher will treat the patients' personal data confidentially and anonymize the data and information in any public release of the results of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR